CLINICAL TRIAL: NCT01654185
Title: Phase II Study of Dimethyldiguanide Combined With AI Compared to AI in Postmenopausal HR(+) Metastatic Breast Cancer.
Brief Title: Dimethyldiguanide Combined With Aromatase Inhibitor (AI) in Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xichun Hu (Other)
Responsible Party: Sponsor-Investigator, Xichun Hu, Deputy director of department of medical oncology, Fudan University
Organization: Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fudan BR2012-12
Record Dates: First submitted 2012-07-27; First posted 2012-07-31 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-01

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole; exemestane; Aromatase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AI plus Dimethyldiguanide (Experimental): AI 1 tablet qd plus Dimethyldiguanide 0.5 bid
  Interventions: Drug: AI plus Dimethyldiguanide
- Aromatase Inhibitor (Active Comparator): AI monotherapy
  Interventions: Drug: Aromatase Inhibitor

INTERVENTIONS:
Drug: AI plus Dimethyldiguanide — AI 1 tablet per day Dimethyldiguanide 0.5 bid
  Other Names: letrozole or exemestane; Dimethyldiguanide
  Arms: AI plus Dimethyldiguanide
Drug: Aromatase Inhibitor — 1 tablet per day
  Other Names: letrozole or exemestane
  Arms: Aromatase Inhibitor

SUMMARY:
The addition of dimethyldiguanide might increase the efficacy of AI treatment in metastatic breast cancer.

DETAILED DESCRIPTION:
The addition of dimethyldiguanide might increase the efficacy of AI in patients with metastatic breast cancer after the failure of the first line endocrine therapy.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal HR positive breast cancer patients;
* inoperable locally advanced or metastatic breast cancer patients;
* candidate for endocrine therapy;
* ECOG equal to or less than 1;
* adequate bone marrow function(Hb>=90g/L, WBC >=3.5×10^9/L,ANC>=1.5×10^9/L, PLT>=80×10^9/L; adequate renal function(Ccr<=ULN);adequate liver function(ALT,AST,AKP<=2.5*ULN,or <=5*ULN if liver metastases)
* life expectancy >=12weeks;
* no severe history disease of liver,heart,lung or kidney;
* written informed consent form;

Exclusion Criteria:

* Her-2 overexpression;
* patients who has visceral endocrisis；

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-07; Primary Completion 2014-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
progression free survival | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Xichun Hu, MD,PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, China